CLINICAL TRIAL: NCT05868317
Title: Induction Chemotherapy With FOLFIRINOX ( 5 Fluorouracil, Oxaliplatine and Irinotecan) Followed by Short Course Radiotherapy in Locally Advanced Rectal Cancer
Brief Title: Induction Chemotherapy Followed by Short Course Radiotherapy in Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Salah Azaïz Cancer Institute (Other)
Responsible Party: Principal Investigator, Amel Mezlini, Professor in Medical Oncology, Salah Azaïz Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISANOX
Record Dates: First submitted 2023-04-14; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer; Locally Advanced
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; folfirinox; Fluorouracil; Oxaliplatin; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction CT followed by short course RT (Experimental): Induction chemotherapy with modified 5 fluorouracil, oxaliplatin and irinotecan followed by short course radiotherapy ( 5x5 Gy), then 5 fluorouracil and oxaliplatin based chemotherapy. Surgery will be performed 6 to 8 weeks after completion of RT.
  Interventions: Drug: Chemotherapy With FOLFIRINOX ( 5 Fluorouracil, Oxaliplatine and Irinotecan); Radiation: Radiotherapy

INTERVENTIONS:
Drug: Chemotherapy With FOLFIRINOX ( 5 Fluorouracil, Oxaliplatine and Irinotecan) — Induction chemotherapy with six cycles of modified 5 fluorouracil,oxaliplatin and irinotecan followed by short course radiotherapy (RT) (5x5 Gy), then two cycles of 5 fluorouracil and oxaliplatin based chemotherapy and surgery will be performed 6 to 8 weeks after completion of RT.
  After surgery , continuation of chemotherapy with 4 cycles of 5 fluorouracil and oxaliplatin regardless of pathological response
Radiation: Radiotherapy — Short Course Radiotherapy

SUMMARY:
A Single-arm phase II trial evaluating induction chemotherapy with FOLFIRINOXm followed by short course radiotherapy (RT) in locally advanced rectal carcinoma

DETAILED DESCRIPTION:
Total neoadjuvant treatment (TNT) is currently the standard of care in the management of locally advanced rectal cancer since recent studies have shown improved pathological complete response and disease-free survival with this approach. However, survival benefits remain unproven.

Two strategies of TNT are validated so far : induction chemotherapy with FOLFIRINOX followed by long course radio-chemotherapy (RCT) or short course RT (5x5 Gy) followed by consolidation chemotherapy with CAPOX (capecitabine and oxaliplatin) or FOLFOX (5 FU and oxaliplatin) .

The objective of investigators is to evaluate pathological complete response with a new strategy of TNT consisting in induction chemotherapy with FOLFIRINOXm followed by short course RT and a delayed surgery.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) performance status : 0 or 1
* Histologically proven rectal adenocarcinoma < 10 cm from anal margin on rectoscopy
* clinically T3 (cT3) or clinically T4 (cT4) and/ or N+ non metastatic rectal cancer
* Neutrophil count > 1500 e/mm3
* Platelet count >100000
* Hemoglobin > 10 g/dl ( transfusion allowed)
* Normal bilirubin level
* Creatinine clearance > 50 ml/mn

Exclusion Criteria:

* Distant metastases
* History of chemotherapy or radiotherapy
* Grade 1 neuropathy
* Patient undergoing treatment for another cancer
* Active infection or severe comorbidities contraindicating chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | 1 month after surgery
  no tumor identified in the rectum or associated lymph nodes by final pathology following surgical resection

SECONDARY OUTCOMES:
Disease free survival | 3 years
  first relapse after surgery
overall survival | 3 years
  death
objective response rate to induction chemotherapy | immediately after completion of 6 cycles of chemotherapy ( each cycle is 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Feryel letaief ksontini, A/Prof, Study Director — Salah Azaiez Institute of oncology; Amina Mokrani, A/Prof, Study Chair — Salah Azaiez Institute; Mouna Ayadi, A/Prof, Study Chair — Salah Azaiez Institute
Locations (1):
- Amel Mezlini, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Fernandez-Martos C, Pericay C, Aparicio J, Salud A, Safont M, Massuti B, Vera R, Escudero P, Maurel J, Marcuello E, Mengual JL, Saigi E, Estevan R, Mira M, Polo S, Hernandez A, Gallen M, Arias F, Serra J, Alonso V. Phase II, randomized study of concomitant chemoradiotherapy followed by surgery and adjuvant capecitabine plus oxaliplatin (CAPOX) compared with induction CAPOX followed by concomitant chemoradiotherapy and surgery in magnetic resonance imaging-defined, locally advanced rectal cancer: Grupo cancer de recto 3 study. J Clin Oncol. 2010 Feb 10;28(5):859-65. doi: 10.1200/JCO.2009.25.8541. Epub 2010 Jan 11. PMID 20065174
- [Result] Conroy T, Bosset JF, Etienne PL, Rio E, Francois E, Mesgouez-Nebout N, Vendrely V, Artignan X, Bouche O, Gargot D, Boige V, Bonichon-Lamichhane N, Louvet C, Morand C, de la Fouchardiere C, Lamfichekh N, Juzyna B, Jouffroy-Zeller C, Rullier E, Marchal F, Gourgou S, Castan F, Borg C; Unicancer Gastrointestinal Group and Partenariat de Recherche en Oncologie Digestive (PRODIGE) Group. Neoadjuvant chemotherapy with FOLFIRINOX and preoperative chemoradiotherapy for patients with locally advanced rectal cancer (UNICANCER-PRODIGE 23): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 May;22(5):702-715. doi: 10.1016/S1470-2045(21)00079-6. Epub 2021 Apr 13. PMID 33862000